CLINICAL TRIAL: NCT04184765
Title: Evaluation of Inflammatory Markers in Laparoscopic and Abdominal Hysterectomies: A Retrospective Study in Kocaeli, Northwest Turkey
Brief Title: Inflammatory Markers in Hysterectomies
Status: Completed | Type: Observational
Sponsor: mehmet ozsurmeli (Other)
Responsible Party: Sponsor-Investigator, mehmet ozsurmeli, medical doctor, Derince Training and Research Hospital
Organization: Derince Training and Research Hospital (Other)
Other Study IDs: 35753575
Record Dates: First submitted 2019-11-27; First posted 2019-12-04 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Gynecologic Disease; Inflammation
Keywords: hysterectomies; inflammation mediators; lymphocyte
MeSH Terms: conditions — Genital Diseases, Female; Inflammation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Maternal venous blood samples were taken into hemogram tubes with 2-2.5 ml ethylenediaminetetraacetic acid (EDTA) and homogenized. The calibrations of the device were completed and analyzed using the Pentra DF Nexus Hematology System® (Horiba Healthcare, Japan). PLR and NLR were calculated by dividing platelet and neutrophil counts, respectively, by the lymphocyte count.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Total laparoscopic hysterectomies: Between 2018 and 2019, data obtained from patients in the LH and AH groups were reviewed retrospectively. The preoperative and postoperative hematocrit (HCT), hemoglobin (HB), white blood cell (WBC), platelet (PLR) and neutrophil-lymphocyte (NLR) ratios and values were compared as well as the demographic characteristics of the patients.
- Abdominal hysterectomies: Between 2018 and 2019, data obtained from patients in the LH and AH groups were reviewed retrospectively. The preoperative and postoperative hematocrit (HCT), hemoglobin (HB), white blood cell (WBC), platelet (PLR) and neutrophil-lymphocyte (NLR) ratios and values were compared as well as the demographic characteristics of the patients.

SUMMARY:
This retrospective study was conducted in the obstetrics and gynecology clinic at Derince Training and Research Hospital.

The study group was identified as patients who underwent hysterectomy between 2018 and 2019. Our hospital is a 50-bed tertiary reference center where approximately 3,500 births per year occur, and about 500 gynecological-oncological surgeries are performed annually. The records of patients who underwent LH and AH were reviewed retrospectively. Preoperative and postoperative blood values in the first 24 hours after surgery were compared: hematocrit (HCT), hemoglobin (HB), WBC, PLR, and NLR values were compared as well as the demographic characteristics of the patients who underwent these procedures. In addition, to evaluate the effect of ovaries on the inflammatory markers, the patients were divided into two groups: oophorectomy and non-oophorectomy.

In our clinic, the decision to perform a hysterectomy is made by the weekly gynecology council. The type of surgery is determined according to the clinical condition of the patient, the gynecological examination, and the patient's request. In general, open surgery is preferred in patients with giant fibroids, many previous surgeries, and immobile uteri. Conditions such as dysfunctional uterine bleeding, cervical intraepithelial neoplasms, and uterine descensus indicate the need for LH. In cases where there is no clinical suspicion, oophorectomy is performed according to the patients' wishes.

In benign cases, the preferred type of hysterectomy is type 1 extra facial hysterectomy. In LH, the procedure is performed as follows: The uterine manipulator is inserted vaginally. First, a Veress needle and then a trocar are entered through the umbilicus. The abdomen is insufflated with carbon dioxide, and the appropriate number of ports is placed. Uterine ligaments and vessels are cut by using bipolar energy. The uterus is removed through the vagina, and the vaginal cuff is sutured laparoscopically.

Patients with chronic diseases (e.g., hypertension, diabetes mellitus, and rheumatologic, nephrological, and hematological diseases), the presence of active infection, corticosteroid use, acetylsalicylic acid, and anticoagulant use were not included in the study. Bladder and bowel injuries, blood transfusion requirements, wound infection and hematoma, postoperative respiratory system complications (e.g., atelectasis) were evaluated as surgical complications.

ELIGIBILITY:
Inclusion Criteria:

* total or abdominal hysterectomy

Exclusion Criteria:

* hypertension, diabetes mellitus, rheumatologic, nephrological, and hematological diseases), the presence of active infection, corticosteroid use, acetylsalicylic acid, and anticoagulant use were not included in the study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: women without any other medical problem who need hysterectomy for any condition
Sampling Method: Non-Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Change of inflammatory markers in abdominal and laparoscopic hysterectomies | 24 hours post-surgery
  Preoperative and postoperative hematocrit (%), hematocrit (%), hemoglobin (gram/deciliter), white blood cell (x103/mm3), PLR, and NLR values values in the first 24 hours after laparoscopic or abdominal hysterectomies were compared.

CONTACTS AND LOCATIONS:
Overall Officials: Ünal Türkay, MD, Study Director — Derince Training and Research Hospital; Bahar Salıcı, MD, Study Chair — Derince Training and Research Hospital; Mehmet Salıcı, MD, Study Chair — Derince Training and Research Hospital; Karanfil Nisan Bölge, MD, Study Chair — Derince Training and Research Hospital
Locations (1):
- Derince Training and Research Hospital, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aarts JW, Nieboer TE, Johnson N, Tavender E, Garry R, Mol BW, Kluivers KB. Surgical approach to hysterectomy for benign gynaecological disease. Cochrane Database Syst Rev. 2015 Aug 12;2015(8):CD003677. doi: 10.1002/14651858.CD003677.pub5. PMID 26264829
- [Background] Allendorf JD, Bessler M, Whelan RL, Trokel M, Laird DA, Terry MB, Treat MR. Postoperative immune function varies inversely with the degree of surgical trauma in a murine model. Surg Endosc. 1997 May;11(5):427-30. doi: 10.1007/s004649900383. PMID 9153168
- [Background] Chapron C, Fauconnier A, Goffinet F, Breart G, Dubuisson JB. Laparoscopic surgery is not inherently dangerous for patients presenting with benign gynaecologic pathology. Results of a meta-analysis. Hum Reprod. 2002 May;17(5):1334-42. doi: 10.1093/humrep/17.5.1334. PMID 11980761
- [Background] Collet D, Vitale GC, Reynolds M, Klar E, Cheadle WG. Peritoneal host defenses are less impaired by laparoscopy than by open operation. Surg Endosc. 1995 Oct;9(10):1059-64. doi: 10.1007/BF00188987. PMID 8553203
- [Background] Cruickshank AM, Fraser WD, Burns HJ, Van Damme J, Shenkin A. Response of serum interleukin-6 in patients undergoing elective surgery of varying severity. Clin Sci (Lond). 1990 Aug;79(2):161-5. doi: 10.1042/cs0790161. PMID 2167805
- [Background] Faist E, Kupper TS, Baker CC, Chaudry IH, Dwyer J, Baue AE. Depression of cellular immunity after major injury. Its association with posttraumatic complications and its reversal with immunomodulation. Arch Surg. 1986 Sep;121(9):1000-5. doi: 10.1001/archsurg.1986.01400090026004. PMID 3741094
- [Background] Fornara P, Doehn C, Seyfarth M, Jocham D. Why is urological laparoscopy minimally invasive? Eur Urol. 2000 Mar;37(3):241-50. doi: 10.1159/000052351. PMID 10720847
- [Background] Gibson PH, Croal BL, Cuthbertson BH, Small GR, Ifezulike AI, Gibson G, Jeffrey RR, Buchan KG, El-Shafei H, Hillis GS. Preoperative neutrophil-lymphocyte ratio and outcome from coronary artery bypass grafting. Am Heart J. 2007 Nov;154(5):995-1002. doi: 10.1016/j.ahj.2007.06.043. PMID 17967611
- [Background] Grace PA, Quereshi A, Coleman J, Keane R, McEntee G, Broe P, Osborne H, Bouchier-Hayes D. Reduced postoperative hospitalization after laparoscopic cholecystectomy. Br J Surg. 1991 Feb;78(2):160-2. doi: 10.1002/bjs.1800780209. PMID 1826624
- [Background] Gupta A, Watson DI. Effect of laparoscopy on immune function. Br J Surg. 2001 Oct;88(10):1296-306. doi: 10.1046/j.0007-1323.2001.01860.x. PMID 11578282
- [Background] Horne BD, Anderson JL, John JM, Weaver A, Bair TL, Jensen KR, Renlund DG, Muhlestein JB; Intermountain Heart Collaborative Study Group. Which white blood cell subtypes predict increased cardiovascular risk? J Am Coll Cardiol. 2005 May 17;45(10):1638-43. doi: 10.1016/j.jacc.2005.02.054. Epub 2005 Apr 25. PMID 15893180
- [Background] Imtiaz F, Shafique K, Mirza SS, Ayoob Z, Vart P, Rao S. Neutrophil lymphocyte ratio as a measure of systemic inflammation in prevalent chronic diseases in Asian population. Int Arch Med. 2012 Jan 26;5(1):2. doi: 10.1186/1755-7682-5-2. PMID 22281066
- [Background] Iwase M, Kondo G, Watanabe H, Takaoka S, Uchida M, Ohashi M, Nagumo M. Regulation of Fas-mediated apoptosis in neutrophils after surgery-induced acute inflammation. J Surg Res. 2006 Jul;134(1):114-23. doi: 10.1016/j.jss.2005.10.013. Epub 2005 Dec 27. PMID 16376940
- [Background] Joris J, Cigarini I, Legrand M, Jacquet N, De Groote D, Franchimont P, Lamy M. Metabolic and respiratory changes after cholecystectomy performed via laparotomy or laparoscopy. Br J Anaesth. 1992 Oct;69(4):341-5. doi: 10.1093/bja/69.4.341. PMID 1419439
- [Background] Khatib G, Soysal C, Cetin C, Gulec UK, Guzel AB, Keskin N, Vardar MA, Gumurdulu D. Does preoperative neutrophil to lymphocyte or platelet to lymphocyte ratios have a role in predicting borderline ovarian tumors? J Ovarian Res. 2016 Nov 8;9(1):78. doi: 10.1186/s13048-016-0283-2. PMID 27821183
- [Background] Kuwae N, Kopple JD, Kalantar-Zadeh K. A low lymphocyte percentage is a predictor of mortality and hospitalization in hemodialysis patients. Clin Nephrol. 2005 Jan;63(1):22-34. doi: 10.5414/cnp63022. PMID 15678693
- [Background] Lennard TW, Shenton BK, Borzotta A, Donnelly PK, White M, Gerrie LM, Proud G, Taylor RM. The influence of surgical operations on components of the human immune system. Br J Surg. 1985 Oct;72(10):771-6. doi: 10.1002/bjs.1800721002. PMID 2412626
- [Background] Malik E, Buchweitz O, Muller-Steinhardt M, Kressin P, Meyhofer-Malik A, Diedrich K. Prospective evaluation of the systemic immune response following abdominal, vaginal, and laparoscopically assisted vaginal hysterectomy. Surg Endosc. 2001 May;15(5):463-6. doi: 10.1007/s004640000348. Epub 2001 Mar 13. PMID 11353962
- [Background] Mealy K, Gallagher H, Barry M, Lennon F, Traynor O, Hyland J. Physiological and metabolic responses to open and laparoscopic cholecystectomy. Br J Surg. 1992 Oct;79(10):1061-4. doi: 10.1002/bjs.1800791024. PMID 1422720
- [Background] Medeiros LR, Stein AT, Fachel J, Garry R, Furness S. Laparoscopy versus laparotomy for benign ovarian tumor: a systematic review and meta-analysis. Int J Gynecol Cancer. 2008 May-Jun;18(3):387-99. doi: 10.1111/j.1525-1438.2007.01045.x. Epub 2007 Aug 10. PMID 17692084
- [Background] Neal CP, Mann CD, Sutton CD, Garcea G, Ong SL, Steward WP, Dennison AR, Berry DP. Evaluation of the prognostic value of systemic inflammation and socioeconomic deprivation in patients with resectable colorectal liver metastases. Eur J Cancer. 2009 Jan;45(1):56-64. doi: 10.1016/j.ejca.2008.08.019. Epub 2008 Oct 9. PMID 18848775
- [Background] Ogawa K, Hirai M, Katsube T, Murayama M, Hamaguchi K, Shimakawa T, Naritake Y, Hosokawa T, Kajiwara T. Suppression of cellular immunity by surgical stress. Surgery. 2000 Mar;127(3):329-36. doi: 10.1067/msy.2000.103498. PMID 10715990
- [Background] Pinto EM, Huppert FA, Morgan K, Mrc Cfas, Brayne C. Neutrophil counts, monocyte counts and cardiovascular disease in the elderly. Exp Gerontol. 2004 Apr;39(4):615-9. doi: 10.1016/j.exger.2003.12.011. PMID 15050297
- [Background] Redmond HP, Watson RW, Houghton T, Condron C, Watson RG, Bouchier-Hayes D. Immune function in patients undergoing open vs laparoscopic cholecystectomy. Arch Surg. 1994 Dec;129(12):1240-6. doi: 10.1001/archsurg.1994.01420360030003. PMID 7986152
- [Background] Sarraf KM, Belcher E, Raevsky E, Nicholson AG, Goldstraw P, Lim E. Neutrophil/lymphocyte ratio and its association with survival after complete resection in non-small cell lung cancer. J Thorac Cardiovasc Surg. 2009 Feb;137(2):425-8. doi: 10.1016/j.jtcvs.2008.05.046. Epub 2008 Aug 29. PMID 19185164
- [Background] Sietses C, Wiezer MJ, Eijsbouts QA, Beelen RH, van Leeuwen PA, von Blomberg BM, Meijer S, Cuesta MA. A prospective randomized study of the systemic immune response after laparoscopic and conventional Nissen fundoplication. Surgery. 1999 Jul;126(1):5-9. doi: 10.1067/msy.1999.98702. PMID 10418585
- [Background] Sietses C, Wiezer MJ, Eijsbouts QA, van Leeuwen PA, Beelen RH, Meijer S, Cuesta MA. The influence of laparoscopic surgery on postoperative polymorphonuclear leukocyte function. Surg Endosc. 2000 Sep;14(9):812-6. doi: 10.1007/s004640010080. PMID 11000359
- [Background] Slade MS, Simmons RL, Yunis E, Greenberg LJ. Immunodepression after major surgery in normal patients. Surgery. 1975 Sep;78(3):363-72. PMID 1098195
- [Background] Szkandera J, Stotz M, Eisner F, Absenger G, Stojakovic T, Samonigg H, Kornprat P, Schaberl-Moser R, Alzoughbi W, Ress AL, Seggewies FS, Gerger A, Hoefler G, Pichler M. External validation of the derived neutrophil to lymphocyte ratio as a prognostic marker on a large cohort of pancreatic cancer patients. PLoS One. 2013 Nov 4;8(11):e78225. doi: 10.1371/journal.pone.0078225. eCollection 2013. PMID 24223776
- [Background] Vaisanen M, Lilius EM, Mustonen L, Raekallio M, Kuusela E, Koivisto M, Vainio O. Effects of ovariohysterectomy on canine blood neutrophil respiratory burst: a chemiluminescence study. Vet Surg. 2004 Sep-Oct;33(5):551-6. doi: 10.1111/j.1532-950X.2004.04077.x. PMID 15362995
- [Background] Walsh SR, Cook EJ, Goulder F, Justin TA, Keeling NJ. Neutrophil-lymphocyte ratio as a prognostic factor in colorectal cancer. J Surg Oncol. 2005 Sep 1;91(3):181-4. doi: 10.1002/jso.20329. PMID 16118772
- [Background] Yamanaka T, Matsumoto S, Teramukai S, Ishiwata R, Nagai Y, Fukushima M. The baseline ratio of neutrophils to lymphocytes is associated with patient prognosis in advanced gastric cancer. Oncology. 2007;73(3-4):215-20. doi: 10.1159/000127412. Epub 2008 Apr 17. PMID 18424885
- [Result] Souza MPA, Lima FMDS, Muniz IP, Pereira IS, Sousa LRO, Galantini MPL, Santos DPD, Figueiredo TB, Silva RAAD. Ovariectomy Modifies TH2, and TH17 Balance in BALB/C Allergic Mice. Iran J Allergy Asthma Immunol. 2017 Dec;16(6):525-536. PMID 29338159
- [Derived] Ozsurmeli M, Turkay U, Salici B, Salici M, Bolge KN, Terzi H. Evaluation of inflammatuar response in hysterectomies: a retrospective study in Kocaeli, Turkey. Ginekol Pol. 2021;92(2):105-109. doi: 10.5603/GP.a2020.0146. Epub 2021 Jan 15. PMID 33448002